CLINICAL TRIAL: NCT04266886
Title: Integration of Self-Hypnosis in an Enhanced Recovery After Surgery (ERAS) Program: A Prospective Randomized Trial
Brief Title: Self-Hypnosis for the Enhanced Recovery After Surgery in Patients With Gynecologic Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0143; NCI-2019-08222 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0143 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-12-30; First posted 2020-02-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Malignant Female Reproductive System Neoplasm; Recurrent Malignant Female Reproductive System Neoplasm; Metastatic Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (usual care) (Active Comparator): Patients receive usual care including receipt of multi-modal analgesia and the injection of a local analgesic at the time of surgery on the ERAS pathway.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (usual care, self-hypnosis guided relaxation) (Experimental): Patients receive usual care as in Arm I. Patients also receive self-hypnosis guided relaxation by listening to MP3 on the ERAS pathway.
  Interventions: Other: Best Practice; Procedure: Hypnotherapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
Procedure: Hypnotherapy — Receive self-hypnosis guided relaxation
  Other Names: Clinical Hypnosis; Hypnosis
  Arms: Arm II (usual care, self-hypnosis guided relaxation)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well self-hypnosis works in enhancing recovery after surgery in patients with gynecologic cancer. A guided relaxation method called self-hypnosis may help affect how patients feel pain and symptoms after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether participation in pre-operative self-hypnosis (SH) is feasible and will improve patients' perception of post-surgical pain, after undergoing open gynecologic surgery (laparotomy) on an enhanced recovery pathway.

SECONDARY OBJECTIVES:

I. To evaluate whether participation in pre-operative SH is associated with changes in use of opioid medication, including time to first postoperative opioid and total dose of opioids taken (converted to morphine equivalents) and avoidance of opioids.

II. To explore whether participation in pre-operative SH is associated with changes in length of stay.

III. To explore whether there are differences between the two study arms in other common symptoms of women undergoing gynecologic surgery, functional recovery after surgery and quality of life (QOL).

IV. To explore whether expectations regarding symptom management or hypnotic susceptibility are related to or influence the perception of symptoms after surgery.

V. To measure satisfaction with the intervention (patients on arm 2). VI. To perform sub analyses to explore whether other common clinical or demographic factors are potential covariates.

EXPLORATORY OBJECTIVE:

I. To compare two different instruments measuring patient reported outcomes in hospital postoperative recovery.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive usual care including receipt of multi-modal analgesia and the injection of a local analgesic at the time of surgery on the enhanced recovery after surgery (ERAS) pathway.

ARM II: Patients receive usual care as in Arm I. Patients also receive self-hypnosis guided relaxation by listening to MP3 on the ERAS pathway.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an exploratory laparotomy for suspected gynecologic cancer, which includes metastatic disease from neoplasia originating in other organs
* Planned participation in the Gynecologic Enhanced Recovery Pathway
* Patient must be able to read, understand, and speak English
* Consents to being part of a randomized study
* Patient has physical and mental capabilities to take part in study

Exclusion Criteria:

* Sensitivity to amide-type local anesthetics
* Patients on long-acting opioid medications, or scheduled (four or more times a day for seven or more days) short-acting opioid medications within the last 30 days
* Emergency surgery of any type that does not allow for proper time for protocol review by the patient
* Surgery that involves known/anticipated resection of anterior abdominal wall with plastic surgery reconstruction
* Patients undergoing known/anticipated anterior abdominal wall hernia repairs
* Patients undergoing pelvic exenteration
* Patients with known major psychiatric disease
* Patients with hearing impairment such that they are unable to hear the intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of participating in pre-operative self-hypnosis | Up to 1 day
  Will assess proportion of participants who listen to the complete audio file in the preoperative holding area.
Patients' perception of post-surgical pain | Post-operative day 1 (POD1)
  Will summarize POD1 pain scores for each treatment arm using descriptive statistics. Will use a Wilcoxon rank sums test to determine if the POD1 pain scores in the self-hypnosis arm are lower than the usual care arm. Pain intensity score from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa A Meyer, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org